CLINICAL TRIAL: NCT01222936
Title: A Phase II Study of the Histone Deacetylase Inhibitor Panobinostat (LBH589) in Patients With Advanced Small Cell Lung Cancer (SCLC)
Brief Title: LBH Phase II in Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Scientific Director, SENDO Tech s.r.l.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S075LBH501
Record Dates: First submitted 2010-10-11; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Small Cell Lung Carcinoma
Keywords: LBH581; Panobinostat; Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: LBH581 — 25 mg/5 ml solution packaged in 6 ml type I glass vials and given as a 30 minutes infusion at the dose of 20 mg/m2 i.v., on day 1 and 8, every 21 days.
  Other Names: Panobinostat

SUMMARY:
SCLC is the most aggressive and lethal form of lung cancer, typically very sensitive to cytotoxic therapy when first diagnosed, but associated with a high incidence of tumour relapse and a very poor life expectancy. Combination chemotherapy based on cisplatin or carboplatin and etoposide represents the most widely used regimen. Despite of the high response rate, approximately 80% of patients with limited disease and nearly all patients with extended disease develop disease relapse or progression. Topotecan is, at present, the only approved second line treatment in Europe.

The search of a new therapeutic agent that could alter the natural history of SCLC would be an important goal to be reached. LBH589 (Panobinostat) is a histone deacetylase (HDAC) inhibitor available for intravenous and oral administration. LBH589 could be classified as PAN-DAC inhibitor targeting both histone and non histone proteins and as such it could be suitable for combination with cytotoxics. Three phase I dose escalation studies with both the intravenous and the oral formulation of LBH589, examining various dose schedules of administration have been conducted in advanced solid tumours and haematological malignancies.

Single agent activity was observed in phase I in patients with haematological cancer. In solid tumours one response (Hormone-refractory Prostatic Cancer) and some prolonged stabilizations have been observed with intravenous formulation. Phase II studies are now in progress.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytological diagnosis of SCLC, mixed small and non small cell tumours are excluded
2. ≤ 2 prior chemotherapy lines
3. Progression after, and not during, last previous chemotherapy treatment
4. Age ≥ 18 and ≤ 75 years
5. Life expectancy of at least 3 months
6. ECOG Performance Status 0-1
7. At least one measurable lesion according to modified RECIST criteria defined as ≥ 1 lesion with longest diameter ≥ 20 mm by conventional techniques or ≥ 10 mm with spiral CT scan. In case of solitary measurable lesion, histological confirmation is not required.
8. Adequate haematological function:

   * haemoglobin ≥ 9 g/dl
   * platelet count ≥ 100,000/mm3
   * neutrophils count ≥ 1,500/mm3
9. Adequate liver and renal functions:

   * Total serum bilirubin ≤ 1.5 x UNL
   * Serum creatinine ≤ 1.5 x UNL or 24 hours creatinine clearance ≥ 50 mL/min
   * AST and ALT ≤ 2.5 x UNL or ≤ 5.0 x UNL if the transaminase elevation is due to hepatic involvement
   * Albumin ≥ 2.5 g/dl
   * Alkaline phosphatase ≤ 2.5 x UNL
10. Fertile patients must use effective contraception during and for ≥ 6 weeks after completion of study therapy
11. Ability to signed informed consent

Exclusion Criteria:

1. Progression while on previous chemotherapy
2. Other chemotherapy treatment < 4 weeks prior to enrolment
3. Presence of active infection
4. A known history of HIV positivity
5. Participation to any investigational drug study < 4 weeks preceding study enrolment
6. Radiotherapy involving > 30% of the active bone marrow
7. Thoracic and brain radiotherapy < 4 weeks prior to enrolment. Palliative radiotherapy is allowed during study treatment
8. Presence of any serious neurological or psychiatric disorder
9. Impaired cardiac function, including any one of the following:

   * Complete Left Bundle Branch Block or obligate use of a cardiac pacemaker or congenital long QT syndrome or history or presence of atrial or ventricular tachyarrhythmias or clinically significant resting bradycardia (< 50 beats per minute) or QTcF > 480 msec on screening ECG or Right Bundle Branch block + left anterior hemiblock (biphasic block)
   * Acute MI ≤ 3 months prior to starting study drug
   * Other clinically significant heart disease (e.g. congestive heart failure, previous history angina pectoris, uncontrolled hypertension, history of labile hypertension or arrhythmia, or history of poor compliance with an antihypertensive regimen)
   * Any other case of current abnormal cardiac functionality or history of cardiac disease causing LVEF < 45% as determined by ECHO
10. Known hypersensitivity/allergic reaction to the study product
11. Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
12. Previous or current concomitant malignancy at other site, other than basal or squamous cell carcinoma of the skin and carcinoma in situ of the uterine cervix, within 3 years.
13. Symptomatic or progressive brain metastases
14. Patients with an active bleeding diathesis or on anticoagulants Therapeutic doses of sodium warfarin (Coumadin) are not allowed. Low doses of Coumadin (e.g., ≤ 2 mg/day) for line patency are allowed
15. Pregnant or lactating women
16. Concomitant use of CYP3A4/5 inhibitors or inducers, or drug that prolong the QT interval and/or induce torsades ventricular arrythmia, where the treatment can not be discontinued or switched to a different medication prior to starting study drug.
17. Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GMCSF) ≤ 2 weeks prior to starting study drug.
18. Unable or unwilling to comply with all study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 12-18 weeks (foreseen participation of the patient in the study)
  Objective response rate measured according to the RECIST (Response Evaluation Criteria In Solid Tumours).

SECONDARY OUTCOMES:
Duration of antitumor activity | 12-18 weeks (foreseen participation of the patient in the study)
  Time-to-progression, duration of response and disease stabilization
Drug safety profile | 28 days following the last dose
  Evaluation of adverse events, physical examination, vital signs, concomitant medications, laboratory (hematology and chemistry) and instrumental data (i.e. ECG) considered for safety analyses

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Marinis, MD, Study Chair — Azienda Ospedaliera San Camillo Forlanini
Locations (8):
- Germany (2):
  - Klinik für Onkologie und Haematologie, Frankfurt am Main
  - Klinikum Kassel Innere Medizin, Kassel
- Italy (6):
  - Azienda Ospedaliera "S. G. Moscati", Avellino, AV
  - Istituto Nazionale Ricerca sul Cancro, Genova, GE
  - U.O. di Oncologia Medica, Palermo, PA
  - Ospedale Maggiore di Parma, Parma, PR
  - Azienda Ospedaliera San Camillo Forlanini, Rome, RM
  - Az. San. Ospedaliera Molinette S. Giovanni Battista di Torino, Torino, TO